CLINICAL TRIAL: NCT04381689
Title: Phase Ⅲ, Randomized, Double-blind, Active Controlled to Evaluate the Immunogenicity and Safety of "IL-YANG Quadrivalent Seasonal Influenza Vaccine" in Healthy Infants From 6 Months to Under 3 Years of Age(≥ 6 Months and < 3 Years)
Brief Title: Phase 3 Study to Evaluate the Immunogenicity and Safety of Inactived Split Influenza Vaccine in Healthy Korea Infants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IF4IC03
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Influenza; Influenza vaccine; Split influenza vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-YANG PFS (Experimental): IL-YANG FLU Vaccine Prefilled Syringe INJ.
  Interventions: Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ.
- GSK PFS (Active Comparator): Fluarix Tetra Pre-filled Syringe
  Interventions: Biological: Fluarix Tetra Pre-filled Syringe

INTERVENTIONS:
Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ. — Teratect Prefilled Syringe Inj. 0.5mL
  Arms: IL-YANG PFS
Biological: Fluarix Tetra Pre-filled Syringe — Fluarix Tetra Pre-filled Syringe 0.5mL
  Arms: GSK PFS

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of IL-YANG Inactivated Split Influenza Vaccine (IL-YANG Quadrivalent Seasonal Influenza Vaccine) in healthy infants from 6 months to under 3 years of age(≥ 6 months and < 3 years)

DETAILED DESCRIPTION:
The study is an Randomized, Double-blind, Active controlled Phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged from 6 months to < 3 years
* Subjects were born after full term pregnancy (37 weeks)
* Voluntary written informed consent was obtained from the subject and the subject's legally acceptable representative (consent of legally acceptable representative was required for subjects younger than 10 years of age (and for subjects younger than 7 years of age for the some institutions)).

Exclusion Criteria:

* Subject with a known allergy to eggs, chicken, neomycin, gentamicin or any components of the study vaccine
* Subject who had received an influenza vaccine within the last 6 months
* Subject who has, or has a family history of, an immune system disorder including immune deficiency disease
* Subject with a history of Guillain-Barre syndrome
* Subject with Down's syndrome or cytogenetic disorders.
* Subject with severe chronic disease which in the investigator's opinion would not make the subject a good candidate for the clinical trial
* Subject with hemophilia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subject who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine
* Subject who had previously received another vaccine within 28 days before administration of the study drug, or is scheduled to receive another vaccine during the study period.
* Subject who had received immunosuppressant or immune modifying drug within the last 3 months prior to administration of the study vaccine
* Subject who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or is expecting to be treated with immunoglobulin or blood-derived products during the study.
* Subject who had participated in another experimental study within 30 days prior to administration of the study vaccine
* Subject with other clinically significant medical or psychological condition who in the investigator's opinion would not be suitable for the study.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate against Hemagglutination Inhibition(HI) antibody | Up to Day28(+7) after the last vaccination
  Seroconversion rate(a lower bound of 95 CI) ≥ 40%
Seroprotection rate against Hemagglutination | Up to Day28(+7) after the last vaccination
  Seroprotection rate(a lower bound of 95 CI) ≥ 70%

SECONDARY OUTCOMES:
Geometric Mean Titer(GMT) | Up to Day28(+7) after the last vaccination
  GMT of HI Antibody Titer Before Vaccination and After Vaccination
Geometric Mean Ratio(GMR) | Up to Day28(+7) after the last vaccination
  GMR of HI Antibody Titer Before Vaccination and After Vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Korea University ANSAN Hospital, Ansan-si, Gyeonnggi-do
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonnggi-do